CLINICAL TRIAL: NCT02301897
Title: A Phase 2, Multi-Center, Parallel Design, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of 6 and 12 mg Proellex® (Telapristone Acetate) Administered Orally in the Treatment of Premenopausal Women With Confirmed Symptomatic Uterine Fibroids
Brief Title: A Multi-Center, Parallel Design, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of 6 and 12 mg Proellex® (Telapristone Acetate) Administered Orally in the Treatment of Premenopausal Women With Confirmed Symptomatic Uterine Fibroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZPU-203
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-05

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Following the baseline assessment no treatment period, matching placebo, orally, once daily for 18 weeks (Treatment Course 1) and repeated for an additional 18 weeks (Treatment Course 2) following the off drug interval (ODI).
  Interventions: Drug: Placebo
- Telapristone Acetate 6 mg (Experimental): Following the baseline assessment no treatment period, telapristone acetate 6 milligrams (mg), orally, once daily for 18 weeks (Treatment Course 1) and repeated for an additional 18 weeks (Treatment Course 2) following the ODI.
  Interventions: Drug: Telapristone Acetate
- Telapristone Acetate 12 mg (Experimental): Following the baseline assessment no treatment period, telapristone acetate 12 mg, orally, once daily for 18 weeks (Treatment Course 1) and repeated for an additional 18 weeks (Treatment Course 2) following the ODI.
  Interventions: Drug: Telapristone Acetate

INTERVENTIONS:
Drug: Telapristone Acetate — Telapristone acetate, orally, once daily for 18 weeks (Course 1) and repeated for an additional 18 weeks (Course 2) following the ODI.
  Other Names: Proellex®
  Arms: Telapristone Acetate 12 mg; Telapristone Acetate 6 mg
Drug: Placebo — Matching placebo, orally, once daily for 18 weeks (Course 1) and repeated for an additional 18 weeks (Course 2) following the ODI.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of two oral doses of Proellex administered for up to 2 courses of treatment (18 weeks each), each separated by an Off-Drug Interval (ODI), to premenopausal women with symptomatic uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Is a pre-menopausal female, between 18 and 47 years
* Participant has a history of at least 3 regular menstrual cycles in which menorrhagia (heavy bleeding) is due to uterine fibroids
* Confirmed uterine fibroid(s) at screening
* Visit 1 historical pictorial blood loss assessment chart of >120 milliliters (mL) of blood loss, to ensure participants have a menstrual blood loss of at least 80 mL by Alkaline Hematin Assay (during the baseline assessment period).
* A Body Mass Index (BMI) between 18 and 45 inclusive

Exclusion Criteria:

* Participant is pregnant or lactating or is attempting or expecting to become pregnant during the entire study period
* Received an investigational drug in the 30 days prior to the screening for this study
* Has an intrauterine device in place
* Observation or history of abnormal endometrial biopsy including the presence of endometrial intraepithelial neoplasia
* Participants with abnormally high liver enzymes or liver disease

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (16):
- United States (16):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Phoenix, Arizona
  - MomDoc Women's Health Research, Scottsdale, Arizona
  - KO Clinical Research, LLC, Fort Lauderdale, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Atlanta Women's Research Institute, Inc., Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Southern Clinical Research Associates, LLC, Metairie, Louisiana
  - Palmetto Clinical Research, Summerville, South Carolina
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - DCT-HCWC, LLC dba Discovery Clinical Trials, Dallas, Texas
  - Advances in Health, Houston, Texas
  - The Women's Hospital of Texas Clinical Research Center, Houston, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Telapristone Acetate 6 mg: Following the baseline assessment no treatment period, telapristone acetate 6 milligrams (mg), orally, once daily for 18 weeks (Treatment Course 1) and repeated for an additional 18 weeks (Treatment Course 2) following the off drug interval (ODI).
- Placebo: Following the baseline assessment no treatment period, matching placebo, orally, once daily for 18 weeks (Treatment Course 1) and repeated for an additional 18 weeks (Treatment Course 2) following the ODI.
Period: Treatment Course 1
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Started | 12 | 17 | 14
Completed | 9 | 14 | 8
Not Completed | 3 | 3 | 6
Not completed — Non-Compliance | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Withdrawal by Sponsor | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Other Miscellaneous Reasons | 1 | 0 | 0
Period: Treatment Course 2
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Started | 9 | 14 | 8
Completed | 8 | 9 | 7
Not Completed | 1 | 5 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Other Miscellaneous Reasons | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who were randomized, received study drug, and had some post-baseline safety data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo | Total
Number analyzed (Participants) | 12 | 17 | 14 | 43
Age, Continuous [Mean (Full Range); unit: years] | 40.8 [31 to 46] | 41.4 [35 to 47] | 41.9 [30 to 47] | 41.4 [30 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 14 | 43
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Amenorrhea at the End of Treatment Course 1
Description: Amenorrhea was defined as no bleeding intensity score greater than 1 using the Daily Diary Card during the 28 days leading up to the last day of dosing at Week 18. Bleeding intensity was graded on a 5-point scale where: 0=no bleeding to 4=heavy bleeding.
Time Frame: At the end of 18-weeks Treatment Course 1
Population: Intent-to-treat (ITT) population consisted of all participants who were randomized and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage of participants | 58.33 | 70.59 | 0.0
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Test type: Superiority; p = 0.0008, Chi-Square Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Test type: Superiority; p < 0.001, Chi-Square Test

2. Secondary Outcome: Percentage of Participants in Amenorrhea at the End of Treatment Course 2
Description: as for outcome 1
Time Frame: At the end of 18-weeks Treatment Course 2
Population: ITT population consisted of all participants who were randomized and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage of participants | 25.00 | 64.71 | 0.0
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Test type: Superiority; p = 0.0719, Chi-Square Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Test type: Superiority; p = 0.0004, Chi-Square Test

3. Secondary Outcome: Change in Pictorial Blood Loss Assessment Chart (PBAC) Score From Baseline to the End of Treatment Courses 1 and 2, ODI Course 1 and the Course 2 Week 28 Follow-up (FU) Visit
Description: Uterine bleeding was assessed with the use of the PBAC, a validated self-reporting method to estimate menstrual blood loss. Participants recorded daily the number of tampons and towels used and the degree to which individual items were soiled with blood (plus small or large clots). Pictorial scores range from score 1 for slightly stained tampon/towel, 5 for a partially stained tampon/towel, 10 for a completely saturated tampon, 20 for a completely saturated towel, and 5 for each episode of flooding and for each blood clot larger than a quarter in size. Total score can range from 0 (no bleeding) to >500. Higher scores indicate more bleeding. Lower scores indicate less bleeding. A negative change from Baseline indicates improvement (reduction in bleeding).
Time Frame: Baseline (No treatment period) to the end of 18-weeks Treatment Course 1, the end of ODI Course 1, the end of 18-weeks Treatment Course 2 and the Course 2 Week 28 FU Visit
Population: ITT population consisted of all participants who were randomized and received study drug. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
score on a scale
  Baseline | 316.82 (162.828) | 371.20 (332.028) | 267.07 (119.334)
  Change from Baseline (CFB) to Week 18 Course 1: number analyzed (Participants) | 10 | 15 | 11
  Change from Baseline (CFB) to Week 18 Course 1 | -340.61 (151.198) | -364.55 (342.572) | -44.48 (468.771)
  CFB to ODI Course 1: number analyzed (Participants) | 12 | 16 | 11
  CFB to ODI Course 1 | -100.92 (238.412) | -127.41 (282.914) | -104.92 (261.137)
  CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 13 | 7
  CFB to Week 18 Course 2 | -323.20 (138.553) | -396.69 (367.242) | -238.86 (164.498)
  CFB to Course 2 Week 28 FU: number analyzed (Participants) | 4 | 3 | 2
  CFB to Course 2 Week 28 FU | -220.50 (137.805) | -655.33 (466.031) | -324.70 (109.884)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; CFB to Week 18 Course 1; Test type: Superiority; p = 0.0167, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; CFB to Week 18 Course 1; Test type: Superiority; p = 0.1257, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; CFB to ODI Course 1; Test type: Superiority; p = 0.9754, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; CFB to ODI Course 1; Test type: Superiority; p = 0.7672, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; CFB to Week 18 Course 2; Test type: Superiority; p = 0.2232, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; CFB to Week 18 Course 2; Test type: Superiority; p = 0.4512, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; CFB to Course 2 Week 28 FU; Test type: Superiority; p = 0.3545, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; CFB to Course 2 Week 28 FU; Test type: Superiority; p = 0.2482, Wilcoxon Rank-Sum Test

4. Secondary Outcome: Percentage Change in PBAC Score From Baseline to the End of Treatment Courses 1 and 2, ODI Course 1 and the Course 2 Week 28 FU Visit
Description: Uterine bleeding was assessed with the use of the PBAC, a validated self-reporting method to estimate menstrual blood loss. Participants recorded daily the number of tampons and towels used and the degree to which individual items were soiled with blood (plus small or large clots). Pictorial scores range from score 1 for slightly stained tampon/towel, 5 for a partially stained tampon/towel, 10 for a completely saturated tampon, 20 for a completely saturated towel, and 5 for each episode of flooding and for each blood clot larger than a quarter in size. Total score can range from 0 (no bleeding) to >500. Higher scores indicate more bleeding. Lower scores indicate less bleeding. A negative percentage change from Baseline indicates improvement (reduction in bleeding).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in PBAC score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in PBAC score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 15 | 11
  Percentage CFB to Week 18 Course 1 | -96.95 (7.952) | -94.58 (16.256) | 59.70 (357.363)
  Percentage CFB to ODI Course 1: number analyzed (Participants) | 12 | 16 | 11
  Percentage CFB to ODI Course 1 | 33.22 (236.393) | 1.41 (85.953) | 6.69 (165.599)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 13 | 7
  Percentage CFB to Week 18 Course 2 | -98.69 (3.448) | -100.00 (0.000) | -75.00 (29.476)
  Percentage CFB to Course 2 Week 28 FU: number analyzed (Participants) | 4 | 3 | 2
  Percentage CFB to Course 2 Week 28 FU | -55.48 (27.739) | -81.59 (20.066) | -99.68 (0.454)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0016, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0003, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to ODI Course 1; Test type: Superiority; p = 0.6666, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to ODI Course 1; Test type: Superiority; p = 0.3612, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0309, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0007, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 28 FU; Test type: Superiority; p = 0.0641, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 28 FU; Test type: Superiority; p = 0.3743, Wilcoxon Rank-Sum Test

5. Secondary Outcome: Percentage Change in Uterine Fibroid System Quality of Life Survey System Severity (UFS-SSS) Score From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. Each question was answered on a 5-point scale where 1=Not at all to 5=A very great deal. The sum of total scores was transformed to a range of 0=no symptoms (best) to 100=most severe symptoms (worst). A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline (No treatment period) to the end of 18-weeks Treatment Course 1, On-drug Course 2, the end of 18-weeks Treatment Course 2 and the Course 2 Week 24 FU Visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 15 | 11
  Percentage CFB to Week 18 Course 1 | -70.41 (14.656) | -68.46 (31.874) | -32.99 (25.658)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 9 | 12 | 8
  Percentage CFB to On-Drug Course 2 | -58.36 (31.193) | -75.40 (28.158) | -44.62 (39.429)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 11 | 7
  Percentage CFB to Week 18 Course 2 | -69.17 (24.150) | -80.23 (29.252) | -56.65 (38.700)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 7 | 9 | 4
  Percentage CFB to Course 2 Week 24 FU | -33.85 (50.603) | -40.45 (42.753) | -60.53 (36.144)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0049, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0064, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.5637, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.0505, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.4262, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.1419, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.4497, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.5371, Wilcoxon Rank-Sum Test

6. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 1 From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 1: During the previous 3 months how distressed were you by "heavy bleeding during your menstrual period"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 15 | 11
  Percentage CFB to Week 18 Course 1 | -87.50 (27.003) | -83.33 (34.932) | -40.91 (39.167)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 9 | 12 | 8
  Percentage CFB to On-Drug Course 2 | -69.44 (37.034) | -95.83 (14.434) | -44.79 (31.477)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 11 | 7
  Percentage CFB to Week 18 Course 2 | -86.11 (28.260) | -95.45 (15.076) | -57.14 (37.401)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 7 | 9 | 4
  Percentage CFB to Course 2 Week 24 FU | -39.29 (31.810) | -25.00 (30.046) | -72.92 (35.600)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0069, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0059, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.2117, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.0006, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0788, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0080, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.1516, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.0565, Wilcoxon Rank-Sum Test

7. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 2 From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 2: During the previous 3 months how distressed were you by "passing blood clots during your menstrual period"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 15 | 11
  Percentage CFB to Week 18 Course 1 | -95.00 (15.811) | -79.44 (41.888) | -40.91 (62.965)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 9 | 12 | 8
  Percentage CFB to On-Drug Course 2 | -66.67 (41.458) | -89.58 (29.113) | -38.54 (45.630)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 11 | 7
  Percentage CFB to Week 18 Course 2 | -80.56 (34.861) | -88.64 (30.339) | -53.57 (50.428)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 7 | 9 | 4
  Percentage CFB to Course 2 Week 24 FU | -54.76 (39.044) | -37.96 (43.123) | -64.58 (41.037)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0110, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0601, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.2168, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.0101, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.2430, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0843, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.5570, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.5302, Wilcoxon Rank-Sum Test

8. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 3 From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 3: During the previous 3 months how distressed were you by "fluctuation in the duration of your menstrual period compared to your previous cycle"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 8 | 14 | 11
  Percentage CFB to Week 18 Course 1 | -65.63 (69.356) | -78.57 (45.844) | -37.88 (35.622)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 8 | 12 | 8
  Percentage CFB to On-Drug Course 2 | -18.75 (134.131) | -56.25 (98.929) | -32.29 (57.466)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 8 | 11 | 7
  Percentage CFB to Week 18 Course 2 | -84.38 (26.517) | -79.55 (60.019) | -55.95 (46.327)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 6 | 9 | 4
  Percentage CFB to Course 2 Week 24 FU | -30.56 (73.156) | -18.52 (103.898) | -25.00 (95.743)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0504, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0151, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.5932, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.0831, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.1416, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0392, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.8275, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.8733, Wilcoxon Rank-Sum Test

9. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 4 From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 4: During the previous 3 months how distressed were you by "fluctuation in the length of your monthly cycle compared to your previous cycles"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 7 | 14 | 10
  Percentage CFB to Week 18 Course 1 | -35.71 (149.204) | -64.29 (65.570) | -15.83 (56.988)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 7 | 11 | 7
  Percentage CFB to On-Drug Course 2 | -14.29 (141.316) | -52.27 (102.746) | 7.14 (103.574)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 7 | 10 | 6
  Percentage CFB to Week 18 Course 2 | -82.14 (27.817) | -77.50 (62.860) | -38.89 (57.413)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 5 | 8 | 3
  Percentage CFB to Course 2 Week 24 FU | -51.67 (38.370) | -45.83 (68.284) | 0.00 (100.000)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0651, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0298, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.4005, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.1114, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.1318, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0807, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.4506, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.4614, Wilcoxon Rank-Sum Test

10. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 5 From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 5: During the previous 3 months how distressed were you by "feeling tightness or pressure in your pelvic area"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 14 | 10
  Percentage CFB to Week 18 Course 1 | -72.50 (24.861) | -76.19 (33.310) | -37.50 (48.631)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 9 | 11 | 8
  Percentage CFB to On-Drug Course 2 | -74.07 (25.154) | -86.36 (30.339) | -56.25 (42.667)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 11 | 7
  Percentage CFB to Week 18 Course 2 | -82.41 (28.396) | -86.36 (30.339) | -64.29 (39.002)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 7 | 9 | 4
  Percentage CFB to Course 2 Week 24 FU | -35.71 (73.396) | -29.63 (41.481) | -58.33 (50.000)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0653, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0480, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.4010, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.0772, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.3206, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.1605, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.5570, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.3437, Wilcoxon Rank-Sum Test

11. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 6 From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 6: During the previous 3 months how distressed were you by "frequent urination during the daytime hours"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 15 | 10
  Percentage CFB to Week 18 Course 1 | -38.33 (39.323) | -46.11 (54.724) | -2.50 (78.572)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 9 | 12 | 7
  Percentage CFB to On-Drug Course 2 | -38.89 (48.591) | -58.33 (63.365) | -61.90 (37.223)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 11 | 6
  Percentage CFB to Week 18 Course 2 | -49.07 (47.952) | -54.55 (65.017) | -34.72 (73.865)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 7 | 9 | 3
  Percentage CFB to Course 2 Week 24 FU | -16.67 (65.793) | -63.89 (48.591) | -80.56 (17.347)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.2624, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0688, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.2790, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.6541, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.8559, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.4326, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.1052, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.9206, Wilcoxon Rank-Sum Test

12. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 7 From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 7: During the previous 3 months how distressed were you by "frequent nighttime urination"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 14 | 9
  Percentage CFB to Week 18 Course 1 | -37.50 (32.691) | -48.81 (47.237) | -18.52 (37.680)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 9 | 11 | 6
  Percentage CFB to On-Drug Course 2 | -43.52 (39.917) | -69.70 (64.039) | -33.33 (52.705)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 10 | 5
  Percentage CFB to Week 18 Course 2 | -32.41 (43.789) | -66.67 (66.667) | -61.67 (43.938)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 7 | 8 | 2
  Percentage CFB to Course 2 Week 24 FU | -27.38 (63.230) | -52.08 (55.946) | -58.33 (11.785)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.1439, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0670, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.6761, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.0639, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.2218, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.4468, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.7678, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.8922, Wilcoxon Rank-Sum Test

13. Secondary Outcome: Percentage Change in the Individual UFS-SSS Subscale Score Question 8 From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Week 24 FU Visit
Description: UFS-SSS is an 8 question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 8: During the previous 3 months how distressed were you by "feeling fatigued"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in UFS-SSS score
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in UFS-SSS score
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 15 | 11
  Percentage CFB to Week 18 Course 1 | -61.67 (21.588) | -58.89 (53.030) | -31.82 (51.750)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 9 | 12 | 8
  Percentage CFB to On-Drug Course 2 | -53.70 (22.864) | -64.58 (41.458) | -43.75 (43.814)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 11 | 7
  Percentage CFB to Week 18 Course 2 | -53.70 (19.145) | -70.45 (37.889) | -53.57 (44.320)
  Percentage CFB to Course 2 Week 24 FU: number analyzed (Participants) | 7 | 9 | 4
  Percentage CFB to Course 2 Week 24 FU | -42.86 (51.015) | -53.70 (35.627) | -56.25 (34.275)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.1262, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.2075, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.5904, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.2430, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.7067, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.2725, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.7016, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Week 24 FU; Test type: Superiority; p = 0.8751, Wilcoxon Rank-Sum Test

14. Secondary Outcome: Percentage Change in Total Uterine Fibroid Volume From Baseline to the End of Treatment Courses 1 and 2, On-drug Course 2 and the Course 2 Off-drug
Description: The total uterine fibroid volume was measured by Magnetic Resonance Imaging (MRI). A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline (No treatment period) to the end of 18-weeks Treatment Course 1, On-drug Course 2, the end of 18-weeks Treatment Course 2 and the Course 2 Off-drug
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in fibroid volume
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
Number analyzed (Participants) | 12 | 17 | 14
percentage change in fibroid volume
  Percentage CFB to Week 18 Course 1: number analyzed (Participants) | 10 | 15 | 9
  Percentage CFB to Week 18 Course 1 | -23.61 (26.553) | -38.91 (20.318) | 1.34 (18.576)
  Percentage CFB to On-Drug Course 2: number analyzed (Participants) | 9 | 12 | 7
  Percentage CFB to On-Drug Course 2 | -29.41 (34.754) | -50.10 (25.048) | 11.88 (56.516)
  Percentage CFB to Week 18 Course 2: number analyzed (Participants) | 9 | 12 | 7
  Percentage CFB to Week 18 Course 2 | -29.41 (34.754) | -50.10 (25.048) | 11.88 (56.516)
  Percentage CFB to Course 2 Off-drug: number analyzed (Participants) | 7 | 9 | 4
  Percentage CFB to Course 2 Off-drug | -31.51 (31.108) | -44.72 (28.406) | -11.26 (37.048)
Statistical Analysis 1: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0338, Wilcoxon Rank-Sum Test
Statistical Analysis 2: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 1; Test type: Superiority; p = 0.0004, Wilcoxon Rank-Sum Test
Statistical Analysis 3: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.0807, Wilcoxon Rank-Sum Test
Statistical Analysis 4: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to On-Drug Course 2; Test type: Superiority; p = 0.0142, Wilcoxon Rank-Sum Test
Statistical Analysis 5: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0807, Wilcoxon Rank-Sum Test
Statistical Analysis 6: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Week 18 Course 2; Test type: Superiority; p = 0.0142, Wilcoxon Rank-Sum Test
Statistical Analysis 7: Comparison: Telapristone Acetate 6 mg vs Placebo; Percentage CFB to Course 2 Off-drug; Test type: Superiority; p = 0.1859, Wilcoxon Rank-Sum Test
Statistical Analysis 8: Comparison: Telapristone Acetate 12 mg vs Placebo; Percentage CFB to Course 2 Off-drug; Test type: Superiority; p = 0.0896, Wilcoxon Rank-Sum Test

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately 46 weeks)
Description: Safety population consisted of all participants who were randomized, received study drug, and had some post-baseline safety data.
Arm/Group | Telapristone Acetate 6 mg | Telapristone Acetate 12 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/17 | 0/14
Other Adverse Events (participants affected / at risk) | 10/12 | 15/17 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telapristone Acetate 6 mg (N=12) | Telapristone Acetate 12 mg (N=17) | Placebo (N=14)
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telapristone Acetate 6 mg (N=12) | Telapristone Acetate 12 mg (N=17) | Placebo (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 4
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Hot flush (General disorders) | 2 | 5 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Lethargy (General disorders) | 0 | 0 | 1
Night sweats (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Asthma (Immune system disorders) | 0 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 2 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 2
Trichomoniasis (Infections and infestations) | 2 | 0 | 2
Fungal infection (Infections and infestations) | 1 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 1 | 0
Dermatitis contact (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0
Weight increased (Investigations) | 1 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Smear cervix abnormal (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 5
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 4 | 8 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 2 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 2 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0
Coital bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
Libido decreased (Reproductive system and breast disorders) | 1 | 0 | 0
Tubo-ovarian abscess (Reproductive system and breast disorders) | 0 | 1 | 0
Vulva cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dizziness (Vascular disorders) | 1 | 1 | 2
Dizziness postural (Vascular disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Vaginal haemorrhage (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT02301897/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT02301897/SAP_001.pdf